CLINICAL TRIAL: NCT05164913
Title: A Retrospective Study of the Effect of General Anesthesia on Children's Behavior
Brief Title: Study of the Effect of General Anesthesia on Children's Behavior
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Other Study IDs: SH9H-2019-T12
Record Dates: First submitted 2021-10-22; First posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-08

CONDITIONS: Behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: No general anesthesia between 0-3 years old or 0-5 years old
  Interventions: Other: Achenbach Child Behavior Checklist （CBCL）scale
- Single anesthesia group: Only once general anesthesia between 0-3 years old or 0-5 years old
  Interventions: Other: Achenbach Child Behavior Checklist （CBCL）scale
- Multiple anesthesia group: More than once general anesthesia between 0-3 years old or 0-5 years old
  Interventions: Other: Achenbach Child Behavior Checklist （CBCL）scale

INTERVENTIONS:
Other: Achenbach Child Behavior Checklist （CBCL）scale — Use the Achenbach Child Behavior Checklist （CBCL）scale to assess children's behavior

SUMMARY:
This topic speculates that there is an interaction between family environment and anesthetic drug exposure on children's behavior. Different family environments have different response to anesthetic drug exposure. Children living in a specific family environment may be more susceptible to the effects of anesthetic drugs. People who are susceptible to exposure to narcotic drugs. In order to clarify this hypothesis and discover specific family environment factors that interact with anesthetic drug exposure, this project intends to establish a retrospective cohort study, through hierarchical analysis and other means, to clarify the behavioral changes of children in different family environments after exposure to anesthetic drugs. Provide theoretical support for the safe application of clinical children's anesthetics.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0-5 who underwent surgery at Shanghai Ninth People's Hospital
* Current age is less than 18 years old
* No surgical complications such as acute infectious diseases, systemic diseases

Exclusion Criteria:

* History of neonatal hypoxic ischemic encephalopathy and bilirubin encephalopathy
* There are genetic diseases or chromosomal diseases, neurological diseases (including epilepsy, congenital diseases), or a history of head trauma, a history of central nervous system infectious diseases, high fever convulsions, congenital heart disease, tumor diseases, and Patients with blood diseases
* People who have autism, attention deficit hyperactivity disorder, or have received behavioral related treatments and interventions
* Those who have undergone cardiovascular surgery, neurosurgery, or those with unstable hemodynamics during surgery
* Those who cannot be contacted, refused to join the group, the questionnaire information does not match the medical records, or the complete medical records cannot be obtained

Ages: 5 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children without basic behavioral abnormalities who have undergone surgery in this hospital
Sampling Method: Non-Probability Sample
Enrollment: 1140 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Achenbach Child Behavior Checklist （CBCL）scale | immediately after the procedure
  sorce（0-100），higher scores mean a worse

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No